CLINICAL TRIAL: NCT05051423
Title: "Mechanisms and Biomarkers of Response and Resistance to Current Targeted Therapies in Gastric Cancer"
Brief Title: "Mechanisms and Biomarkers of Response and Resistance to Current Targeted Therapies in Gastric Cancer" (THERRES)
Acronym: THERRES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy Craiova (Other)
Collaborators: Institutul Clinic Fundeni (Other)
Responsible Party: Sponsor
Other Study IDs: THERRES
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; perfusion pattern in gastric cancer; CHI-EUS
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endosonography; Gastroscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood samples; biopsy samples of normal and gastric cancer tissue;
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with primary gastric tumors referred to our department for EUS local staging.: Patients will be included or excluded according to the following criteria used throughout the study:
  * Inclusion criteria: Patients diagnosed with primary gastric tumors referred for local staging by EUS (n=40); Age 18 to 90 years old, men or women; Signed informed consent for EUS with contrast-enhancement and tissue sampling
  * Exclusion criteria: Prior treatment with chemo-radiotherapy; Failure to provide informed consent; severe coagulopathy.
  Data collected for each participant will include: Personal data (name, surname, age, sex); results from previous investigations (blood count, liver and renal function tests, tumoral markers, gastroscopy, computed tomography), EUS variables (including CEH-EUS), histological and immunohistochemical findings, TNM and pTNM status (if possible), molecular analysis findings.
  Interventions: Diagnostic Test: Endoscopic ultrasound

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound — Imaging tests:
  All patients will be evaluated by EUS and CEH-EUS, using radial EUS instruments. Prior to the investigation the stomach has to be empty for at least 8 hours. During the examination biopsies will be taken from normal and tumor tissue for gene expression analysis.
  CEH-EUS procedure:
  A two panel image with the usual conventional gray-scale B-mode EUS image on the right side and with the contrast harmonic image on the left side will be used, according to pre-established presets. The starting point of the timer will be considered the moment of intravenous contrast injection (Sonovue 2,4 mL), with the whole movie (T0-T120s) recorded on the embedded HDD of the ultrasound system for later analysis
  Molecular tests:
  Blood analysis. Whole blood (1ml) will be collected before imaging procedures in an Eppendorf tube on EDTA solution.
  Biopsy samples of normal and GC tissue. Gene expression will be analyzed using qPCR with Taqman®- labeled probes.
  Other Names: Upper endoscopy; Blood sampling

SUMMARY:
The main aim was to assess the tumor vascular perfusion pattern in gastric cancer (GC). The investigators used dynamic contrast harmonic imaging endoscopic ultrasound (CHI-EUS) and the results were compared with the immunohistochemical expression of CD105 and clinico-pathological parameters.

DETAILED DESCRIPTION:
The study design is prospective and will include patients with gastric tumors referred to Gastroenterology Department from University of Medicine and Pharmacy of Craiova for EUS local staging enrolled during 18 months.

Data collected for each participant will include: Personal data (name, surname, age, sex); results from previous investigations (blood count, liver and renal function tests, tumoral markers, gastroscopy, computed tomography), EUS variables (including CEH-EUS), histological and immunohistochemical findings, TNM and pTNM status (if possible), molecular analysis findings.

Imaging tests All patients will be evaluated by EUS and CEH-EUS, using radial EUS instruments. Prior to the investigation the stomach has to be empty for at least 8 hours. During the examination biopsies will be taken from normal and tumor tissue for gene expression analysis. For EUS examination, the patient will be placed in left lateral position. The EUS scope will be inserted under direct vision, passed by the tumor and examination should begin during withdrawal at 7.5 MHz. The tumor will be characterized describing its echogenicity, echostructure, size, extent into the wall and surrounding structures, and it will be staged using the modification of the TNM classification. The presence/absence of power Doppler signals will be noted. All lymph nodes will be reported with their maximal size, echogenicity, shape and margins. Nodes larger than 5 mm in diameter, with hypoechoic appearance, round shape (rather than ovoid or flat), sharply demarcated borders and located nearby the tumor will be suspected for malignancy.

CEH-EUS procedure: A two panel image with the usual conventional gray-scale B-mode EUS image on the right side and with the contrast harmonic image on the left side will be used, according to pre-established presets. The examination will be performed at a low mechanical index (dynamic wide-band contrast harmonic imaging mode) of 0.2. The starting point of the timer will be considered the moment of intravenous contrast injection (SonoVue 2,4 mL), with the whole movie (T0-T120s) recorded on the embedded HDD of the ultrasound system for later analysis. Parameters for objective measurement of tumor perfusion will include maximum intensity of enhancement, mean transit time, time to peak (wash-in time), wash-in slope, area under the curve, representing indirectly blood flow or blood volume in GC patients.

Complications may occur during EUS, but they are rare. These consist of bleeding at the biopsy site which is usually minimal, self-limited and rarely requires follow-up. Perforation of the stomach is extremely rare. The safety profile of the ultrasound contrast agent (Sonovue®) showed a very low incidence of side effects. It is not nephrotoxic and the incidence of hypersensitivity or severe allergic events is lower than with current X-ray agents and comparable to that of other magnetic resonance contrast agents. Sono-Vue is approved for clinical use in EU countries.

The biological material collected during the study will be frozen and stored. This will include one ml of whole blood and 4 tissue biopsies (2 from normal tissue and 2 from the tumour) of 2 to 3 mm each. When the expected number of participants is reached, the samples will undergo molecular studies for assessing the markers of angiogenesis as detailed further in the protocol. The biological materials will be stored and analysed during an estimated time of 20 months from the start of the trial. Biopsy samples for immunohistochemistry will be included in formalin solution and sent at pathology laboratory.

Molecular tests

* Blood analysis. Whole blood (1ml) will be collected before imaging procedures in an Eppendorf tube on EDTA solution, placed immediately at 40C for maximum 24 hours, and then kept at - 800C for later analysis of angiogenic factors.
* Biopsy samples of normal and GC tissue. Gene expression will be analyzed using qPCR with Taqman®- labeled probes. To quantify the results obtained by real-time RT-PCR the standard curve method will be used. The paired-samples will be collected in RNAlater (Ambion), stored at 40C for 12- 24 hours, and then kept at - 800C. Later analysis will assess the genes expression of angiogenic markers.

Immunohistochemistry IHC will be focused of angiogenic markers: VEGF-A family and their receptors: VEGFR as well as tyrosine kinases receptors (RTKs).

The VEGF-C expression in tumor samples (marker of lymphangiogenesis) will be quantified. Furthermore, a correlation between EUS findings (N stage) and VEGF-C expression will be established.

The microvessel density (MVD) will be calculated using immunohistochemistry for CD105.

Statistical analysis The estimated number of participants enrolled to the study is at least 50 during first 24 months. Both descriptive data analysis and statistical inference will be performed.

Correlations between CE-EUS parameters and pathologic and genetic findings will be analyzed using the T-test and the Pearson correlation coefficient (r) for continuous data, while the Chi-square test will be applied for categorical data. One-way analysis of variance (ANOVA) will be performed for comparison between different subgroups (T stages). Survival analysis from the moment of diagnosis will be evaluated using Kaplan-Meyer curves. Traditional parameters as TNM stage, type of treatment will be analyzed. Statistical significance will be defined as a p-value less than 0.05.

These minimal risks will be outweighed by the potential implications for future patient care.

Research subjects will receive consent on behalf of written and oral information before inclusion in the study. The interview will cover detailed information, including an understandable presentation of the project with its predictable risks and side-effects, expected outcomes and benefits from the research.

Any unplanned events or adverse effects will be reported immediately to the Regional Ethics Committee on biomedical research.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with primary gastric adenocarcinoma;
* no neoadjuvant therapy;
* age: 18 to 90 years old;
* gender: men or women;
* signed informed consent for EUS with contrast-enhancement and tissue sampling;

Exclusion Criteria:

* other types of gastric cancer than adenocarcinoma;
* prior treatment with chemo-radiotherapy;
* failure to provide informed consent;
* severe coagulopathy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with primary gastric tumors referred for local staging by EUS; Age 18 to 90 years old, men or women;
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Correlations with statistical significance between time-intensity curve analysis parameters, immunohistochemical markers of angiogenesis and clinico-pathological parameters. | 1 year
  The investigators expect to see correlations with statistical significance between immunohistochemical markers of angiogenesis (CD105), clinico-pathological and time-intensity curve (TIC) parameters :peak enhancement (PE), wash-in area under the curve (WiAUC), rise time (RT), mean transit time (mTTI), time to peak (TTP), wash-in rate (WiR), wash-in perfusion index (WiPI), wash-outAUC (WoAUC) and wash-in and wash-outAUC (WiWoAUC), fall time (FT), wash-out rate (WoR), quality of fit (QOF), region of interest area (ROI area).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center in Gastroenterology and Hepatology, University of Medicine and Pharmacy, Craiova, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folkman J. Fundamental concepts of the angiogenic process. Curr Mol Med. 2003 Nov;3(7):643-51. doi: 10.2174/1566524033479465. PMID 14601638
- [Background] Kerbel RS. Tumor angiogenesis. N Engl J Med. 2008 May 8;358(19):2039-49. doi: 10.1056/NEJMra0706596. No abstract available. PMID 18463380
- [Background] Shibuya M, Claesson-Welsh L. Signal transduction by VEGF receptors in regulation of angiogenesis and lymphangiogenesis. Exp Cell Res. 2006 Mar 10;312(5):549-60. doi: 10.1016/j.yexcr.2005.11.012. Epub 2005 Dec 5. PMID 16336962
- [Background] Smith NR, Baker D, James NH, Ratcliffe K, Jenkins M, Ashton SE, Sproat G, Swann R, Gray N, Ryan A, Jurgensmeier JM, Womack C. Vascular endothelial growth factor receptors VEGFR-2 and VEGFR-3 are localized primarily to the vasculature in human primary solid cancers. Clin Cancer Res. 2010 Jul 15;16(14):3548-61. doi: 10.1158/1078-0432.CCR-09-2797. Epub 2010 Jul 6. PMID 20606037
- [Background] Li L, Wang L, Song P, Geng X, Liang X, Zhou M, Wang Y, Chen C, Jia J, Zeng J. Critical role of histone demethylase RBP2 in human gastric cancer angiogenesis. Mol Cancer. 2014 Apr 9;13:81. doi: 10.1186/1476-4598-13-81. PMID 24716659
- [Background] Ferrara N. Vascular endothelial growth factor. Eur J Cancer. 1996 Dec;32A(14):2413-22. doi: 10.1016/s0959-8049(96)00387-5. No abstract available. PMID 9059329
- [Background] Ulyatt C, Walker J, Ponnambalam S. Hypoxia differentially regulates VEGFR1 and VEGFR2 levels and alters intracellular signaling and cell migration in endothelial cells. Biochem Biophys Res Commun. 2011 Jan 21;404(3):774-9. doi: 10.1016/j.bbrc.2010.12.057. Epub 2010 Dec 17. PMID 21168388
- [Background] Chen CN, Hsieh FJ, Cheng YM, Cheng WF, Su YN, Chang KJ, Lee PH. The significance of placenta growth factor in angiogenesis and clinical outcome of human gastric cancer. Cancer Lett. 2004 Sep 15;213(1):73-82. doi: 10.1016/j.canlet.2004.05.020. PMID 15312686
- [Background] Kondo K, Kaneko T, Baba M, Konno H. VEGF-C and VEGF-A synergistically enhance lymph node metastasis of gastric cancer. Biol Pharm Bull. 2007 Apr;30(4):633-7. doi: 10.1248/bpb.30.633. PMID 17409493
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768